CLINICAL TRIAL: NCT00070928
Title: Polysomnographic Assessment of Alternative Treatments for Sleep Disturbance in Parkinson's Disease
Brief Title: Valerian to Improve Sleep in Patients With Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01AT000611-01 (NIH)
Record Dates: First submitted 2003-10-09; First posted 2003-10-13 (Estimated); Last update posted 2006-07-26 (Estimated); Status verified 2006-07

CONDITIONS: Insomnia; Parkinson's Disease
Keywords: Sleep
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Parkinson Disease | interventions — Valeriana extract

INTERVENTIONS:
Drug: valerian

SUMMARY:
The purpose of this trial is to test the short-term effectiveness of valerian, a medicinal herb, to improve sleep in patients with Parkinson's disease (PD).

DETAILED DESCRIPTION:
Patients with PD have exceptionally poor sleep. Sleep in patients with PD is characterized by excessive activity in surface electromyographic (EMG) recordings from many different muscle groups. Despite sleep disturbances, approximately 50% of patients experience a transient (1 to 3 hour) reduction in waking motor symptoms upon arising in the morning. This effect has been termed Sleep Benefit. This study will evaluate the effects of valerian, a medicinal herb, on the sleep of patients with PD.

This is a 17 day study where participants will be evaluated by polysomnography on days one, two, three, sixteen and seventeen.. Polysomnographic measurements will include customary variables such as total sleep time, sleep efficiency, and sleep latency, as well as EMG measures of periodic and isolated muscle activity during sleep. Participants will be required to keep a detailed sleep log of their self reported sleep characteristics across the entire 17 study nights. Outcomes will include measures of both nocturnal sleep and waking motor function. Assessments of motor function will be made the morning immediately following Nights 3 and 17 in order to test for improvement related to improved sleep. On the morning following Night 17, participants are provided with a one-week supply of valerian in an Open Label extension. Participants are provided an additional Sleep Log for this week and asked to return the Sleep Log when they complete the Open Label phase.

ELIGIBILITY:
Inclusion Criteria

* Idiopathic Parkinson's disease
* Willing to undergo overnight, in-lab polysomnography
* Sufficient literacy to allow completion of sleep logs
* Stable doses and timing of all Parkinsonian medications during the course of the trial

Exclusion Criteria

* Dementia
* Parkinsonism secondary to toxic, infectious, or other medical conditions
* History of stroke, cerebellar disease, or progressive supranuclear palsy
* History of liver or renal disease
* History of duodenal or bladder obstruction

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2000-09; Study Completion 2006-06

CONTACTS AND LOCATIONS:
Overall Officials: Donald L. Bliwise, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University Medical School/Wesley Woods Hospital, Atlanta, Georgia, United States